CLINICAL TRIAL: NCT02881086
Title: Treatment Optimization in Adult Patients With Newly Diagnosed Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma by Individualised, Targeted and Intensified Treatment - a Phase IV-trial With a Phase III-part to Evaluate Safety and Efficacy of Nelarabine in T-ALL Patients
Brief Title: Optimization of Therapy in Adult Patients With Newly Diagnosed Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma by Individualised, Targeted and Intensified Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, GMALL Head, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMALL08_2013
Record Dates: First submitted 2016-08-04; First posted 2016-08-26 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: Acute lymphoblastic leukemia; Lymphoblastic lymphoma; Nelarabine; BCR-ABL; MRD; PEG-Asparaginase; Rituximab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Rituximab; nelarabine; pegaspargase; Cranial Irradiation; Imatinib Mesylate; Idarubicin; Dexamethasone; Cyclophosphamide; fludarabine; Vincristine; Mercaptopurine; Etoposide; Daunorubicin; Methotrexate; Stem Cell Transplantation; Cytarabine; Vindesine; Doxorubicin; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Stratification I - Standard Risk (SR)/ High Risk (HR) (Other): Induction and consolidation I therapy for standard and high risk patients, PH/BCR-ABL-negative Chemotherapy, immunotherapy, intrathecal prophylaxis, CNS irradiation according to randomisation I Drugs: Rituximab, Vincristine, Daunorubicin, Dexamethasone, Cyclophosphamide, Cytarabine, Mercaptopurine, PEG-Asparaginase, Methotrexate, Vindesine, VP16
  Interventions: Drug: Rituximab; Drug: PEG-Asparaginase; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Mercaptopurine; Drug: VP16; Drug: Daunorubicin (DNR); Drug: Methotrexate; Drug: Cytarabine; Drug: Vindesine
- Stratification I - Philadelphia (PH)+ (Other): Induction and consolidation I therapy for PH+ patients Chemotherapy, immunotherapy, intrathecal prophylaxis Drugs: Rituximab, Vincristine, Imatinib, Dexamethasone, PEG-Asparaginase, Cytarabine, Methotrexate, Vindesine, VP16
  Interventions: Drug: Rituximab; Drug: PEG-Asparaginase; Drug: Imatinib; Drug: Dexamethasone; Drug: Vincristine; Drug: VP16; Drug: Methotrexate; Drug: Cytarabine; Drug: Vindesine
- Rand I - B-Lin + CNS Rad + i.th. MTX (Active Comparator): Chemotherapy according to Stratification I SR/HR CNS prophylaxis: CNS irradiation 24 Gy, intrathecal Methotrexate
  Interventions: Procedure: Cranial irradiation; Drug: Methotrexate
- Rand I - B-Lin + i.th. MTX (Experimental): Chemotherapy according to Stratification I SR/HR CNS prophylaxis: intrathecal Methotrexate
  Interventions: Drug: Methotrexate
- Stratification II - SR + MRD-neg (Other): Chemotherapy, immunotherapy, intrathecal prophylaxis, consolidation II, reinduction, consolidation III - VI, maintenance Drugs: Rituximab, PEG-Asparaginase, Cytarabine, Methotrexate, Vindesine, Adriamycin, Prednisolone, Cyclophosphamide, Nelarabine, Dexamethasone
  Interventions: Drug: Rituximab; Drug: Nelarabine; Drug: PEG-Asparaginase; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Cytarabine; Drug: Vindesine; Drug: Adriamycin; Drug: Prednisolone
- Stratification II - HR + MRD-neg (Other): Chemotherapy or stem cell transplantation according to randomisation II
  Interventions: Drug: Rituximab; Drug: Nelarabine; Drug: PEG-Asparaginase; Drug: Cyclophosphamide; Drug: Methotrexate; Procedure: Stem cell transplantation; Drug: Cytarabine; Drug: Vindesine; Drug: Adriamycin; Drug: Prednisolone
- Stratification II - SR/HR/PH+ + MRD-pos (Other): Chemotherapy or targeted therapy, followed by stem cell transplantation Drugs: Fludarabine, Idarubicin, Cytarabine, Nelarabine
  Interventions: Drug: Nelarabine; Drug: Idarubicin; Drug: Fludarabine; Drug: Cytarabine
- Randomisation II - HR + MRD-neg-SCT (Active Comparator): Stem cell transplantation
  Interventions: Procedure: Stem cell transplantation
- Randomisation II - HR + MRD-neg-SR-chemo (Experimental): Chemotherapy, immunotherapy, intrathecal prophylaxis, consolidation II, reinduction, consolidation III - VI, maintenance Drugs: Rituximab, Dexamethasone, PEG-Asparaginase, Cytarabine, Methotrexate, Vindesine, Adriamycin, Prednisolone, Cyclophosphamide, Nelarabine
  Interventions: Drug: Rituximab; Drug: Nelarabine; Drug: PEG-Asparaginase; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Cytarabine; Drug: Vindesine; Drug: Adriamycin; Drug: Prednisolone

INTERVENTIONS:
Drug: Rituximab
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR); Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg
Drug: Nelarabine
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg; Stratification II - SR/HR/PH+ + MRD-pos
Drug: PEG-Asparaginase
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR); Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg
Procedure: Cranial irradiation
  Arms: Rand I - B-Lin + CNS Rad + i.th. MTX
Drug: Imatinib
  Arms: Stratification I - Philadelphia (PH)+
Drug: Idarubicin
  Arms: Stratification II - SR/HR/PH+ + MRD-pos
Drug: Dexamethasone
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR); Stratification II - SR + MRD-neg
Drug: Cyclophosphamide
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification I - Standard Risk (SR)/ High Risk (HR); Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg
Drug: Fludarabine
  Arms: Stratification II - SR/HR/PH+ + MRD-pos
Drug: Vincristine
  Arms: Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR)
Drug: Mercaptopurine
  Arms: Stratification I - Standard Risk (SR)/ High Risk (HR)
Drug: VP16
  Arms: Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR)
Drug: Daunorubicin (DNR)
  Arms: Stratification I - Standard Risk (SR)/ High Risk (HR)
Drug: Methotrexate
  Arms: Rand I - B-Lin + CNS Rad + i.th. MTX; Rand I - B-Lin + i.th. MTX; Randomisation II - HR + MRD-neg-SR-chemo; Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR); Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg
Procedure: Stem cell transplantation
  Arms: Randomisation II - HR + MRD-neg-SCT; Stratification II - HR + MRD-neg
Drug: Cytarabine
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR); Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg; Stratification II - SR/HR/PH+ + MRD-pos
Drug: Vindesine
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification I - Philadelphia (PH)+; Stratification I - Standard Risk (SR)/ High Risk (HR); Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg
Drug: Adriamycin
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg
Drug: Prednisolone
  Arms: Randomisation II - HR + MRD-neg-SR-chemo; Stratification II - HR + MRD-neg; Stratification II - SR + MRD-neg

SUMMARY:
A phase IV study with the primary goal to optimize therapy of adult patients with acute lymphoblastic leukemia or lymphoblastic lymphoma (LBL) by dose and time intensive, pediatric based chemotherapy, risk adapted stem cell transplantation (SCT) and minimal residual disease (MRD) based individualised and intensified therapy. Study will further evaluate the role of asparaginase intensification, the extended use of rituximab and the use of nelarabine as consolidation therapy in T-ALL in a phase III-part of the study. Furthermore two randomisations will focus on the role of central nervous system (CNS) irradiation in combination with intrathecal therapy versus intrathecal therapy only in B-precursor ALL/LBL and the role of SCT in high-risk patients with molecular complete remission. Finally a new, dose reduced induction therapy in combination with Imatinib will be evaluated in Ph/BCR-ABL positive ALL.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia (pro-B, common, pre-B, early T, thymic T, mature T)
* Lymphoblastic lymphoma (B or T-lineage)
* Age 18-55 yrs
* Written informed consent
* Adequate contraception as specified per protocol

Exclusion Criteria:

* Severe comorbidity or leukemia associated complications
* Late relapse of pediatric ALL or ALL as second malignancy
* Cytostatic pre-treatment
* Pregnancy or breast feeding
* Severe psychiatric illness or other circumstances which may compromise cooperation of the patient
* Participation in other clinical trials interfering with the study therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1023 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Event free survival | 3.5 years

SECONDARY OUTCOMES:
Time until consolidation treatment I | approximately 70 days
Disease free survival | 1 year

OTHER OUTCOMES:
Hematological remission rate | after induction, approximately 6-8 weeks from diagnosis
Molecular remission rate | after induction and consolidation, approximately 6-8 weeks from diagnosis
Results of the positron emission tomography (PET) based remission evaluation | after consolidation, approximately 8-10 weeks
Remission duration | up to 10 years
Relapse rate | up to 10 years
Overall survival | up to 10 years
Relapse location | at timepoint of relapse (up to 10 years)
Early death | during induction, approximately 6-8 weeks from diagnosis
Death in clinical remission (CR) | during treatment, up to approximately 2.5 years from diagnosis
Comorbidities according to Charlson Score | up to 2.5 years
Quality of life assessed by QLQ-C30 | up to 2.5 years
Eastern Cooperative Oncology Group (ECOG) under therapy | up to 2.5 years
Toxicity assessed by CTCAE v4.03 | up to 2.5 years
Results of the Dementia Detection (DemTect) test | up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Gökbuget, Dr. med., Principal Investigator — University Hospital of Frankfurt (Main)
Locations (1):
- University Hospital of Frankfurt (Main), Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No